# Short, Online Child Behavior Support Program Study Provider Consent Form

You are invited to be in a research study to learn if a short, online child behavior support program can help kids and their parents. You are being invited because you are a medical provider at a Hennepin Healthcare Clinic. You are one of about 35 medical providers being asked to be in this study. This study is being done by a University of Minnesota team led by Chris Mehus, PhD. Funds for this study are being provided by the National Institute Of Mental Health (NIMH).

### What would I be asked to do?

You would receive a referral process and online directory of therapists who can provide GenerationPMTO, an evidence-based child behavior support program. Half of participating providers will receive a 60-90 minute inperson training in the referral process and how to effectively motivate parents during the referral. The other half of participating providers will receive a written description of the referral process. Over the next year, any time that you provided services to a family that met the screening criteria, you would refer the parents to a therapist who can provide GenerationPMTO.

You would also be asked to fill out an online questionnaire after you review the referral process and after the pilot study year. Each questionnaire will take about 30 minutes. In the questionnaire, we will ask about your background and the acceptability, appropriateness, and feasibility of the referral process and communication skill straining. After you complete each questionnaire, you will be given a \$50 gift card as a thank you for your time and effort.

We would ask Hennepin Healthcare for the total number of clients age 3-5 you saw during the pilot year and the total number of referrals you made.

After the pilot year, you would be invited to a focus group. You will be asked to meet online with a research team member and 5-12 of the other providers participating in this study. The research team member will ask questions to the group about how you liked the referral process, including what was useful and not useful. The meeting will be audio-recorded and will take 90 minutes. After you have completed the focus group, you will be given a \$100 gift card as a thank you for your time and effort.

### Are there risks in being in this study?

There are no major risks to you. You may find some of the questions hard to answer. There is a small risk of loss of privacy. You don't have to answer any questions that you don't want to answer. There is also a small risk of frustration, stress, or sense of added burden by study activities.

# Are there benefits of being in this study?

We cannot promise any benefits to you or others from your taking part in this research. We hope the ability to make a referral for moderate concerns will increase appointment efficiency as well as increase access to child behavior supports. We aim to make this referral process a smooth and simple part of primary care visits that reduces provider load. If you are assigned to the communication skills training, you may learn new tips and strategies for supporting and motivating clients.

This study may benefit others, by making effective parenting programs and referral systems more accessible to families of kids with behavior challenges.

Version Date: <Date>

## What about privacy?

The records of this study are private. Your responses will not be shared with your healthcare providers. Study participants' names will **never** be used in any report of this study. All study records will be kept locked. Only the researchers will have access to study records.

# What if I don't want to be in this study?

That is OK. The study's research team wants to be sure that no one feels pressured to be in the study. If you do decide to be in this study, you can withdraw at any time. Your decision whether or not to participate will not affect your current or future relations with your health care providers or the University of Minnesota.

# What if I have further questions?

Printed Name of Person Obtaining Consent

signed document.

If you have any questions, **you are encouraged** to contact Chris Mehus at 651-785-3660 or email <a href="mailto:cjmehus@umn.edu">cjmehus@umn.edu</a>. Any feedback you have is welcome and provides valuable insight to the research team.

To share feedback privately with the HRPP about your research experience, call the Research Participants' Advocate Line at 612- 625-1650 (Toll Free: 1-888-224-8636) or go to z.umn.edu/participants

Your signature documents your permission to take part in this research. You will be provided a copy of this

| Signature of Participant Printed Name of Participant | Date<br> |
|-------------------------------------------------------|----------|